CLINICAL TRIAL: NCT03357939
Title: A Phase 1 Randomized,Double-Blind and Parallel Controlled Single-dose Clinical Trial of Pharmacokinetics, Safety, Tolerability and Immunogenicity of HLX03 Compared With Humira® From China Source in Chinese Healthy Male Subjects
Brief Title: Phase I Study of HLX3 vs Adalimumab in Chinese Healthy Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Shanghai Henlius Biotech (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: HLX03-HV01
Record Dates: First submitted 2017-11-26; First posted 2017-11-30 (Actual); Last update posted 2022-05-09 (Actual); Status verified 2022-05

CONDITIONS: Immune System Disorder
Keywords: HLX03; adalimumab; pharmacokinetics; biosimilar
MeSH Terms: conditions — Immune System Diseases | interventions — adalimumab biosimilar HS016; Adalimumab

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- HLX03 (Experimental): There are about 68 subjects in this group will receive a single dose of 40 mg of HLX03 in 0.8 mL in subcutaneous injection.
  Interventions: Drug: HLX03
- Humira (Active Comparator): There are about 68 subjects in this group will receive a single dose of 40 mg of Humira in a pre-filled syringe in subcutaneous injection.
  Interventions: Drug: adalimumab

INTERVENTIONS:
Drug: HLX03 — A single dose of 40 mg HLX03 in 0.8 mL in subcutaneous injection.
  Other Names: adalimumab biosimilar
  Arms: HLX03
Drug: adalimumab — A single dose of 40 mg Humira in 0.8 mL in a pre-filled syringe
  Other Names: Humira
  Arms: Humira

SUMMARY:
This healthy male volunteers study will evaluate 148 subjects who will receive a single sub-cutaneous dose of HLX03 （a monoclonal antibody against TNF-a, 40 mg/ 0.8 mL） or Adalimumab(Humira,China spourced,40 mg/0.8 mL injection with a single-use prefilled syringe). This study will involve sampling,pharmacokinetics, safety, tolerability and immunogenicity evaluation of drug levels following administration of HLX03 and the licensed adalimumab products.

DETAILED DESCRIPTION:
This is a randomized, doubl-blinded, parellel-controlled phase 1 PK, safety, tolerability and immunogenicitiy study to compare HLX03, designed as an Adalimumab biosimilar, with China sourced Humira in Chinese health volunteers. All enrolled subjects will receive a single dose of HLX03 (40 mg）or Humira(adalimumab, 40 mg) in subcutaneous injectioin after randomization.

The purpose of this study to prove the similarity in PK, Safety, tolerability and immunogenicity beween HLX03（adalimumab biosimilar） and China sourced Humira and provide evidence for Phase III comparison study.

The blood will be collected before drug administration, and at 1 hr、4 hr、8 hr、24 hr (1d)、48 hr (2d)、72 hr (3d)、96 hr (4d)、、144 hr (6d)、192 hr (8d)、240 hr (10d)、 336 hr (14d)、504 hr (21d)、672 hr (28d)、840 hr (35d)、1008 hr (42d)、1176 hr (49d)、1344 hr (56d)、1680 hr (70d) after drug injection for PK, ADA, etc analysis. All subjects also will be followed up at 0, 1,2,3,4,6,8,10,14,21,28,35, 42, 49, 56, and 70 days after drug administration for AE and other specified outcomes.

The main endpoint is AUC from time zero to ∞. The second endpoints include Cmax, Tmax, T1/2, CL, Vd and AUC（0-last）.

This is single center study in China.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy Chinese males (age: 18~45 yrs) with contraception during and 3 months post-dose. Healthy is defined as no clinically relevant abnormalities identified by a detailed medical history, full physical examination including blood pressure, pulse, ECG, and laboratory testing.
2. BMI between 19.0 and 28.0 kg/m² and body weight between 55 kg and 80 kg.

Exclusion Criteria:

1. suffering from active or latent tuberculosis or history of tuberculosis;
2. have heart disease or a history of heart disease;
3. suffer from mental illness or psychiatric history;
4. suffering from malignant tumors and their history;
5. suffering from herpes zoster and its history;
6. suffering from epilepsy and history of epilepsy;
7. be allergic to the drugs or its components with high sensitivity or allergic reaction, detection of ADA (+);
8. patients who lost blood or donated more than 200 mL within the first 2 months before the screening;
9. major surgery performed within 30 days prior to signing ICF;
10. live vaccine inoculation or vaccination within 12 weeks of screening, or possible administration of vaccine during screening and study visits;
11. previous application of adalimumab or its biosimilars, or anti-TNF alpha drugs;
12. participating in other clinical trials within the first 3 months of the trial;
13. abnormal immune function within 4 weeks before screening;
14. the presence of invasive systemic fungal infection or other opportunistic infections within 2 months prior to screening;
15. systemic or local infection, such as the risk of sepsis and / or known active inflammation within 2 months before screening;
16. 2 months before the screening, there were severe infections in the hospital and / or the need for intravenous antibiotics;
17. 4 or more upper respiratory tract infections occurred within 6 months prior to randomization;
18. hepatitis B surface antigen (HBsAg) positive; if hepatitis B surface antigen (HBsAg) negative, hepatitis B core antibody (HBcAb) positive, peripheral blood hepatitis B virus deoxyribonucleic acid (DNA) test >0 IU/ml also ruled out;
19. hepatitis C virus (HCV) antibody positive;
20. human immunodeficiency virus (HIV) antibody positive;
21. Treponema pallidum (Treponema pallidum, TP) antibody positive;
22. anti nuclear antibody titer was 1:100 examination;
23. drug abusers, alcohol addicts;
24. , the researchers discretion of failure to follow the requirements of the program, instructions and research limitations, such as uncooperative attitude, unable to return to the Research Center for follow-up visits, or unable to complete the entire clinical study.

Ages: 18 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 220 (Actual)
Dates: Start 2017-01-12 (Actual); Primary Completion 2018-09-15 (Actual); Study Completion 2018-09-15 (Actual)

PRIMARY OUTCOMES:
Maximum Concentration（Cmax） of Adalimumab After Single SC Injection of HLX03/Humira | 71 days post-dose
Area Under the Plasma Concentration-time Curve From Zero (0) Hours to the last quantifiable concentration | 71 days post-dose

SECONDARY OUTCOMES:
Area Under the Plasma Concentration-time Curve From Zero (0) to Time Infinity | 71 days post-dose
Time to Maximum Concentration（Tmax） of Adalimumab After Single SC Injection | 71 days post-dose
Half-life time of adalimumab after single SC injection of HXL03/Humira | 71 days

CONTACTS AND LOCATIONS:
Overall Officials: Yanhua Ding, MD, Principal Investigator — The 1st affiliated hospital, Jilin University, PRC
Locations (1):
- the 1st affiliated hospital of Jilin University, Changchun, Jilin, China

REFERENCES:
- [Result] Zhang H, Wu M, Sun J, Zhu X, Li C, Ding Y, Zhang X, Chai K, Li X. Pharmacokinetics, safety, and immunogenicity of HLX03, an adalimumab biosimilar, compared with reference biologic in healthy Chinese male volunteers: Results of a randomized, double-blind, parallel-controlled, phase 1 study. Pharmacol Res Perspect. 2021 Apr;9(2):e00733. doi: 10.1002/prp2.733. PMID 33682358
- See also: FRI0086 CHINA-MANUFACTURED ADALIMUMAB BIOSIMILAR, HLX03, DEMONSTRATED PHARMACOKINETIC EQUIVALENCE AND COMPARABLE SAFETY TO REFERENCE ADALIMUMAB，EULAR 2019 (Poster); Annals of the Rheumatic Diseases — http://dx.doi.org/10.1136/annrheumdis-2019-eular.1909